CLINICAL TRIAL: NCT06021145
Title: Effectiveness of Empagliflozin Added to Automated Insulin Delivery (AID) Systems in Adults With Type 1 Diabetes With Sub-optimal Glycemic Outcomes: a Randomized Controlled Parallel Trial
Brief Title: Effectiveness of Empagliflozin Added to Automated Insulin Delivery (AID) Systems in Adults With Type 1 Diabetes With Sub-optimal Glycemic Outcomes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Diabetes Canada (Other)
Responsible Party: Principal Investigator, Melissa-Rosina Pasqua, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-9953
Record Dates: First submitted 2023-08-21; First posted 2023-09-01 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; empagliflozin; 26-week
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 2.5 mg daily (Experimental): Empagliflozin is a sodium/glucose cotransporter 2 inhibitor (SGLT2i) that inhibits glucose reabsorption in the kidney. In this study, a capsule of empagliflozin 2.5 mg will be taken daily in conjunction with the participant's personal automated insulin delivery system for 26 weeks.
  Interventions: Drug: Empagliflozin
- Placebo (Active Comparator): As a control, a placebo capsule will be taken daily in conjunction with the participant's personal automated insulin delivery system for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — 26-week use of automated insulin delivery system with empagliflozin (2.5 mg daily) in individuals with suboptimal time in range.
  Arms: Empagliflozin 2.5 mg daily
Drug: Placebo — 26-week use of automated insulin delivery system with placebo (daily) in individuals with suboptimal time in range.
  Arms: Placebo

SUMMARY:
The goal of this 26-week multicenter, randomized, parallel, placebo-controlled trial is to test the effectiveness of empagliflozin use in conjunction with automated insulin delivery (AID) to improve glucose control in individuals with type 1 diabetes who do not meet target recommendations for time in range (3.9-10.0 mmol/L). The main question it aims to answer is:

- Will use of empagliflozin (2.5 mg/day) increase time spent in the target range of 3.9 to 10.0 mmol/L compared to placebo for individuals on an AID system who do not meet glycemic targets?

Participants will either take 2.5 mg of empagliflozin or a placebo daily for 26 weeks while remaining on their current AID system.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years of age.
* A clinical diagnosis of type 1 diabetes for at least one year, as per the investigators' clinical judgment (confirmatory C-peptide and antibodies will not be required).
* Minimum 3-month use of a commercial advanced AID system.
* Time in range (3.9 to 10.0 mmol/L) < 70% on their personal AID system in the 30 days prior to screening (with minimum 70% time spent in closed-loop mode).
* Agreement to use a highly effective method of birth control for individuals of child-bearing age and active avoidance of pregnancy during the trial. Child-bearing potential refers to participants of the female sex post-menarche who have not reached menopause and who do not have a disclosed medical condition causing sterility (ex: hysterectomy). Post-menopausal state refers to the absence of menses for 12 months without any alternative cause.

Exclusion Criteria:

* Current or ≤ 2 week use of any anti-hyperglycemic agent other than insulin (such as SGTL2i).
* Current or ≤ 1 month use of Glucagon-like Peptide 1 (GLP1)-Receptor Agonists.
* Current or ≤ 1 month use of supraphysiological doses of oral or intravenous glucocorticoids.
* Planned or ongoing very low carbohydrate diet (< 50g/day).
* Glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 as per CKD-EPI formula with creatinine levels measured within the last 12 months.
* Use of hydroxyurea.
* Planned or ongoing pregnancy.
* Breastfeeding.
* Ongoing active risk of recurrent genito-urinary infections, as per the clinical judgement of the investigators.
* Severe hypoglycemic episode within 1 month of screening, defined as an event resulting in seizure, loss of consciousness, or need to present to the emergency department.
* Diabetic ketoacidosis within 6 months of screening, defined as an event requiring the need to present to medical attention and administration of intravenous insulin.
* Any serious medical illness likely to interfere with the ability to complete the trial per the judgment of the investigators.
* Clinically significant retinopathy as judged by the investigator.
* Recent (< 3 months) acute macrovascular event (ex: acute coronary syndrome or cardiac surgery).
* Prior serious reaction to SGLT2i.
* Use of the Medtronic 670G or 770G system in the last 30 days.
* In the opinion of the investigator, inability to observe the contraindications of the study drugs, or failure to comply to the study protocol or research team's recommendations (e.g., changing pump parameters, ketone measurements).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of time of glucose levels spent in the target range (empagliflozin vs placebo) | 4 weeks
  Target range is defined to be between 3.9 and 10.0 mmol/L of placebo on an automated insulin delivery system vs empagliflozin (2.5 mg) on an automated insulin delivery system. Percent measured as per continuous glucose monitor (CGM) data.

SECONDARY OUTCOMES:
Percentage of time spent in the glucose range between 3.9 and 7.8 mmol/L | 4 weeks
  Percent as per CGM data
Percentage of time spent in the glucose range below 3.9 mmol/L and 3.0 mmol/L | 4 weeks
  Percent as per CGM data
Percentage of time spent in the glucose range above 10.0 mmol/L and 13.9 mmol/L | 4 weeks
  Percent as per CGM data
Mean glucose levels | 4 weeks
  Defined as per CGM data, in mmol/L
Standard deviation of glucose levels | 4 weeks
  Defined as per CGM data, in mmol/L
Coefficient of variance of glucose levels | 4 weeks
  Percent as per CGM data
Total insulin delivery (overall, basal, and bolus) | 4 weeks
  Defined as per participant's pump data
Mean daily carbohydrate intake | 4 weeks
  Defined as per participant's pump data
HbA1c | 26 weeks
  Percent as per blood test
Estimated glomerular filtration rate (eGFR) | 26 weeks
  mL/min/1.73 m^2 as per blood test
Lipid profile | 26 weeks
  Includes measurements in mmol/L as per blood test: total cholesterol, triglycerides, HDL-C, LDL-C, nonHDL-C
Brain Natriuretic Peptide (NT-pro-BNP) | 26 weeks
  ng/L as per blood test
Liver profile - bilirubin | 26 weeks
  umol/L as per blood test
Liver profile - alanine transaminase (ALT) and alkaline phosphatase (ALP) | 26 weeks
  U/L as per blood test
Measurement of body mass: weight and height | 26 weeks
  Body measurement as described (weight in kilograms and height in meters). Weight and height will be combined to report body mass index in kg/m^2.
Waist and hip circumference, and waist-to-hip ratio | 26 weeks
  Body measurements as described (waist and hip circumference in centimeters). Waist and hip cirumference will be combined to report waist-to-hip ratio.
Heart rate | 26 weeks
  Body measurement as described (beats per minutes)
Blood pressure | 26 weeks
  Body measurement as described (diastolic and systolic pressure; mmHg)
Average scores between interventions based on Type 1 Diabetes Distress Scale Questionnaire | 26 weeks
  Self-report scale (1 min = "not a problem" to 6 max = "a very serious problem") that assesses a participant's distress surrounding their diabetes with higher scores correlating to higher distress.
Average scores between interventions based on Hypoglycemic Fear Survey - II | 26 weeks
  Likert scale (1 min to 5 max) that assesses a participant's worry surrounding hypoglycemia with higher scores indicating increased fear of hypoglycemia.
Average scores between interventions based on Diabetes Treatment Satisfaction Questionnaire | 26 weeks
  Self-report scale (0 min = "very dissatisfied" to 6 max = "very satisfied") that assesses a participant's satisfaction surrounding the treatment for their diabetes with higher scores indicating greater satisfaction with treatment.
Fasting ketone levels | 7 days
  As per ketone test strip and meter; measured by participant

CONTACTS AND LOCATIONS:
Overall Officials: Melissa-Rosina Pasqua, MD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The raw data (that is, insulin delivery, glucose levels and individual participant data) and informed consent form will be shared by the corresponding author, for academic purposes, subject to a material transfer agreement and approval of the McGill University Health Center's Research Ethics Board. All data shared will be de-identified. Raw data will be shared for non-commercial use upon reasonable request and a material transfer agreement.
Supporting Information: ICF